CLINICAL TRIAL: NCT02273973
Title: A Phase II Randomized, Double-Blind Study of Neoadjuvant Letrozole Plus GDC-0032 Versus Letrozole Plus Placebo in Postmenopausal Women With ER-positive/HER2-negative, Early Stage Breast Cancer
Brief Title: A Study of Neoadjuvant Letrozole + Taselisib Versus Letrozole + Placebo in Post-Menopausal Women With Breast Cancer (LORELEI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: SOLTI Breast Cancer Research Group (Other); Breast International Group (Other); Austrian Breast and Colorectal Cancer Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GO28888; 2013-000568-28 (EudraCT Number)
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Results first posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; 2-(3-(2-(1-isopropyl-3-methyl-1H-1,2-4-triazol-5-yl)-5,6-dihydrobenzo(f)imidazo(1,2-d)(1,4)oxazepin-9-yl)-1H-pyrazol-1-yl)-2-methylpropanamide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Letrozole + Placebo (Placebo Comparator): Participants will receive 2.5 mg letrozole tablets orally QD along with placebo on a 5-days-on/2-days-off schedule for a total of 16 weeks.
  Interventions: Drug: Letrozole; Other: Placebo
- Letrozole + Taselisib (Experimental): Participants will receive 2.5 milligrams (mg) letrozole tablets orally once daily (QD) along with taselisib tablets at 4 mg (two 2 mg tablets) orally on a 5 days-on/2 days-off schedule for a total of 16 weeks.
  Interventions: Drug: Letrozole; Drug: Taselisib

INTERVENTIONS:
Drug: Letrozole — Letrozole tablets will be administered orally at 2.5 mg QD for 16 weeks.
Other: Placebo — Placebo tablets matched to taselisib formulation will be administered orally daily on 5 days-on/2 days-off schedule for up to 16 weeks.
  Arms: Letrozole + Placebo
Drug: Taselisib — Taselisib will be administered orally at 4 mg (two 2 mg tablets) daily.
  Other Names: GDC-0032
  Arms: Letrozole + Taselisib

SUMMARY:
This is a two-arm, randomized, double-blind, multicenter, pre-operative study to evaluate the effect of combining letrozole and GDC-0032 (also known as taselisib) versus letrozole and placebo in postmenopausal women with estrogen receptor-positive (ER+)/human epidermal growth factor receptor 2 (HER2) untreated, Stage I-III operable breast cancer. Participants will be randomized into one of the two treatment arms with a 1:1 randomization ratio. Letrozole at 2.5 milligrams (mg) will be dosed once daily plus either Taselisib at 4 mg (two 2-mg tablets) or placebo on a 5 days-on/ 2 days-off schedule for a total of 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female participants
* Postmenopausal status
* Histologically confirmed invasive breast carcinoma, with all of the following characteristics: (i) Primary tumor greater than or equal to (>/=) 2 centimeters (cm) in largest diameter (cT1-3) by MRI; (ii) Stage I to operable Stage III breast cancer; (iii) Documented absence of distant metastases (M0)
* Estrogen receptor-positive (ER+) and human epidermal growth factor receptor 2-negative (HER2-) breast cancer
* Breast cancer eligible for primary surgery
* Tumor tissue from formalin-fixed paraffin-embedded cores (FFPE) core biopsy of breast primary tumor that is confirmed as evaluable for phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA) mutation status by central histopathology laboratory
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Fasting glucose less than or equal to (</=) 125 milligrams per deciliter (mg/dL)
* Adequate hematological, renal, and hepatic function
* Absence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Ability and willingness to comply with study visits, treatment, testing, and to comply with the protocol, in the investigator's judgment

Exclusion Criteria:

* Any prior treatment for primary invasive breast cancer
* Participants with cT4 or cN3 stage breast tumors
* Bilateral invasive, multicentric, or metastatic breast cancer
* Participants who have undergone excisional biopsy of primary tumor and/or axillary lymph nodes or sentinel lymph node biopsy
* Type 1 or 2 diabetes requiring antihyperglycemic medication
* Inability or unwillingness to swallow pills
* Malabsorption syndrome or other condition that would interfere with enteric absorption
* History of prior or currently active small or large intestine inflammation (such as Crohn's disease or ulcerative colitis). Any predisposition for gastrointestinal (GI) toxicity requires prior approval from the Medical Monitor.
* Congenital long QT syndrome or QT interval corrected using Fridericia's formula (QTcF) >470 milliseconds (msec)
* Diffusing capacity of the lungs for carbon monoxide (DLCO) <60% of the predicted values
* Clinically significant (i.e., active) cardiovascular disease, uncontrolled hypertension, unstable angina, history of myocardial infarction, cardiac failure class II-IV
* Any contraindication to MRI examination
* Active infection requiring intravenous antibiotics
* Participants requiring any daily supplemental oxygen
* Clinically significant history of liver disease, including viral or other known hepatitis, current alcohol abuse, or cirrhosis
* Any other diseases, active or uncontrolled pulmonary dysfunction, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, that may affect the interpretation of the results, or renders the participants at high risk from treatment complications
* Significant traumatic injury within 3 weeks prior to initiation of study treatment
* Major surgical procedure within 4 weeks prior to initiation of study treatment
* Inability to comply with study and follow-up procedures
* History of other malignancy within 5 years prior to screening, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (117):
- United States (8):
  - Breastlink Med Group Inc, Santa Ana, California
  - MGH Cancer Center, Boston, Massachusetts
  - MSKCC at Basking Ridge, Basking Ridge, New Jersey
  - MSKCC @ Commack, Commack, New York
  - MSKCC @ West Harrison, Harrison, New York
  - Memorial Sloan-Kettering Cancer Center; Hematology/Oncology, New York, New York
  - MSKC @ Rockville, Rockville Centre, New York
  - MD Anderson Cancer Center, Houston, Texas
- Australia (5):
  - Kinghorn Cancer Centre; St Vincents Hospital, Darlinghurst, New South Wales
  - Newcastle Mater Misericordiae Hospital; Oncology, Waratah, New South Wales
  - Victorian Breast and Oncology Care, East Melbourne, Victoria
  - Cabrini Medical Centre; Oncology, Malvern, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (10):
  - Lkh-Univ. Klinikum Graz; Klinik Für Gynäkologie, Graz
  - LKH-UNIV. KLINIKUM GRAZ; Klinische Abteilung für Onkologie, Graz
  - Tiroler Landeskrankenanstalten Ges.M.B.H.; Abt. Für Gynäkologie, Innsbruck
  - Ordensklinikum Linz Barmherzige Schwestern ; Abt. f. Allgemein- und Viszeralchirurgie, Linz
  - Brustzentrum - Ordination Dr. Wette, Saint Veit/Glan
  - Lkh Salzburg - Univ. Klinikum Salzburg; Iii. Medizinische Abt., Salzburg
  - Medizinische Universität Wien; Univ.Klinik für Chirurgie - Abt. für Allgemeinchirurgie, Vienna
  - Medizinische Universität Wien; Univ.Klinik für Frauenheilkunde - Klinik für Gynäkologie, Vienna
  - Krankenhaus Der Stadt Wien-Hietzing; Abt. Für Gynäkologie U. Geburtshilfe, Vienna
  - Klinikum Kreuzschwestern Wels; Iii. Interne Abt., Wels
- Belgium (5):
  - Institut Jules Bordet, Brussels
  - CHU Brugmann (Victor Horta), Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Antwerpen, Edegem
  - Clinique Ste-Elisabeth, Namur
- Brazil (5):
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Instituto Brasileiro De Controle Do Câncer - IBCC; Laboratório De Patologia, São Paulo, São Paulo
- Hospital Clinico Vina del Mar, Viña del Mar, Chile
- Czechia (4):
  - Fakultni Nemocnice Hradec Kralove; Dept of Radiotherapy & Oncology, Hradec Králové
  - Fakultni nemocnice Olomouc; Onkologicka klinika, Olomouc
  - MULTISCAN, s.r.o., Radiologicke centrum Pardubice, Pardubice
  - Oblastni nemocnice Pribram, Příbram
- Hospital Oncologia; Oncology, San Salvador, El Salvador
- France (7):
  - Centre Jean Perrin; Division De Recherche Clinique, Clermont-Ferrand
  - Centre Jean Bernard, Le Mans
  - Institut Curie; Oncologie Medicale, Paris
  - Hopital Saint Louis; Service Onco Thoracique, Paris
  - Centre Rene Huguenin; ONCOLOGIE GENETIQUE, Saint-Cloud
  - CHI de Toulon - Hôpital Sainte Musse, Toulon
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
- Germany (13):
  - Praxisklinik Krebsheilkunde für Frauen / Brustzentrum (Dres. Kittel/Klare), Berlin
  - Studienzentrum Berlin City, Berlin
  - Onkologische Schwerpunktpraxis Bielefeld, Bielefeld
  - Universitätsklinikum "Carl Gustav Carus" der Technischen Universität Dresden, Dresden
  - Klinikum Essen-Mitte Ev. Huyssens-Stiftung / Knappschafts GmbH; Klinik für Senologie / Brustzentrum, Essen
  - Evangelische Kliniken Gelsenkirchen GmbH; Brustzentrum, Gelsenkirchen
  - Universitätsklinikum Hamburg-Eppendorf (UKE); Klinik und Poliklinik für Gynäkologie, Hamburg
  - Medizinische Hochschule Hannover, Klinik für Frauenheilkunde und Geburtshilfe, Hanover
  - Universitätsklinikum Schleswig-Holstein / Campus Lübeck; Klinik für Frauenheilkunde und Geburtshilfe, Lübeck
  - Rotkreuzklinikum München; Frauenklinik, München
  - Universitätsklinikum Münster; Klinik für Frauenheilkunde und Geburtshilfe, Münster
  - Universitätsklinikum Ulm Am Michelsberg; Frauenklinik, Ulm
  - Marien-Hospital Witten; Frauenklinik Brustzentrum, Witten
- Guatemala (2):
  - Centro Oncológico Sixtino / Centro Oncológico SA, Guatemala City
  - Grupo Angeles, Guatemala City
- Hungary (5):
  - Szent Margit Hospital; Dept. of Oncology, Budapest
  - Debreceni Egyetem, Klinikai Kozpont, Onkologiai Klinika, Debrecen
  - Bacs-Kiskun Megyei Korhaz, SZTE AOK Oktato Korhaza, Onkoradiologiai Kozpont, Kecskemét
  - B-A-Z County Hospital, Miskolc
  - Szegedi Tudomanyegyetem, AOK, Szent-Gyorgyi Albert Klinikai Kozpont, Onkoterapias Klinika, Szeged
- Italy (7):
  - Azienda Ospedaliero-Universitaria S.Orsola-Malpighi; Unità Operativa Oncologia Medica, Bologna, Emilia-Romagna
  - Ospedale degli Infermi, Rimini, Emilia-Romagna
  - Uni Degli Studi Di Genova ; Clinica Di Medicina Interna Ad Indirizzo Oncologico, Genoa, Liguria
  - ASST DI CREMONA; Dip. Medicina - S.C. Oncologia, Cremona, Lombardy
  - Ospedale Per Acuti Mater Salutis Di Legnago, Legnago, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 1, Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO); Ricerca Di Senologia Medica, Milan, Lombardy
- Mexico (3):
  - Centro Estatal de Cancerología, Chihuahua City
  - Instituto Nacional De Cancerologia; Oncology; Tumores Mamarios, Distrito Federal
  - Consultorio de Medicina Especializada; Dentro de Condominio San Francisco, Mexico City
- Centro Oncologico America, Panama City, Panama
- Peru (3):
  - Hospital Nacional Cayetano Heredia; Hematology - Oncology, Lima
  - Oncosalud Sac; Oncología, Lima
  - Clinica Internacional, Sede San Borja; Unidad de Investigacion de Clínica Internacional, Lima
- Poland (6):
  - Centrum Onkologii;Im. Franciszka Lukaszczyka;Onkologii, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii i Radioterapii, Gdansk
  - Wojewódzki Szpital Specjalistyczny im. M. Kopernika; Oddział Chemioterapii, Lodz
  - Europejskie Centrum Zdrowia Otwock Szpital im. Fryderyka Chopina, Klinika Onkologii, Otwock
  - Wielkopolskie Centrum Onkologii; im. Marii Skłodowskiej-Curie, Poznan
  - Cent.Onkologii-Instytut im. M. S-Curie, Klinika Now. Piersi i Chirurgii Rekon, Warsaw
- Portugal (3):
  - IPO de Lisboa; Servico de Oncologia Medica, Lisbon
  - Centro Clinico Champalimaud; Oncologia Medica, Lisbon
  - IPO do Porto; Servico de Oncologia Medica, Porto
- South Korea (4):
  - National Cancer Center; Medical Oncology, Gyeonggi-do
  - Seoul National Uni Hospital; Dept. of Internal Medicine/Hematology/Oncology, Seoul
  - Yonsei University Severance Hospital; Medical Oncology, Seoul
  - Samsung Medical Centre; Division of Hematology/Oncology, Seoul
- Spain (17):
  - Hospital Provincial de Castellon; Servicio de Oncologia, Castellon, Castellon
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Servicio de Oncologia, Santiago de Compostela, LA Coruña
  - Instituto Universitario Dexeus; Servicio de Oncología, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital San Pedro De Alcantara; Servicio de Oncologia, Cáceres
  - Hospital Universitari de Girona Dr. Josep Trueta; Servicio de Oncologia, Girona
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico; Servicio de Oncologia, Jaén
  - Hospital Universitari Arnau de Vilanova de Lleida; Servicio de Oncologia, Lleida
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Centro Integral Oncologico Clara Campal (CIOCC); Dirección Médica, Madrid
  - Hospital Universitario de Fuenlabrada; Servicio de Oncologia, Madrid
  - Hospital Universitario Virgen del Rocio; Servicio de Oncologia, Seville
  - Hospital Clinico Universitario; Oncologia, Valencia
  - Hospital Arnau de Vilanova (Valencia) Servicio de Oncologia, Valencia
  - Fundación IVO, Valencia
- Switzerland (3):
  - Kantonsspital Baden; Frauenklinik, Baden
  - Kantonsspital Graubünden;Onkologie und Hämatologie, Chur
  - Fondazione Oncologia Lago Maggiore, Locarno
- United Kingdom (4):
  - Royal Bournemouth General Hospital; Oncology, Bournemouth
  - Frimley Park Hospital; Breast Resaerch Team, Camberley
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Christie Hospital, Manchester

REFERENCES:
- [Derived] Eiger D, Brandao M, de Azambuja E. Lessons learned at SABCS 2019 and to-dos from immunotherapy in breast cancer. ESMO Open. 2020 Mar;5(2):e000688. doi: 10.1136/esmoopen-2020-000688. No abstract available. PMID 32188717
- [Derived] Eiger D, Franzoi MA, Ponde N, Brandao M, de Angelis C, Schmitt Nogueira M, de Hemptinne Q, de Azambuja E. Cardiotoxicity of trastuzumab given for 12 months compared to shorter treatment periods: a systematic review and meta-analysis of six clinical trials. ESMO Open. 2020 Feb;5(1):e000659. doi: 10.1136/esmoopen-2019-000659. PMID 32079624
- [Derived] Saura C, Hlauschek D, Oliveira M, Zardavas D, Jallitsch-Halper A, de la Pena L, Nuciforo P, Ballestrero A, Dubsky P, Lombard JM, Vuylsteke P, Castaneda CA, Colleoni M, Santos Borges G, Ciruelos E, Fornier M, Boer K, Bardia A, Wilson TR, Stout TJ, Hsu JY, Shi Y, Piccart M, Gnant M, Baselga J, de Azambuja E. Neoadjuvant letrozole plus taselisib versus letrozole plus placebo in postmenopausal women with oestrogen receptor-positive, HER2-negative, early-stage breast cancer (LORELEI): a multicentre, randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Oncol. 2019 Sep;20(9):1226-1238. doi: 10.1016/S1470-2045(19)30334-1. Epub 2019 Aug 8. PMID 31402321

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited post-menopausal participants with breast cancer in 22 countries from November 2014 to March 2017.
Groups:
- Experimental: Taselisib + Letrozole: Participants received 2.5 milligrams (mg) letrozole tablets orally once daily (QD) along with taselisib tablets at 4 mg (two 2 mg tablets) orally on a 5 days-on/2 days-off schedule for a total of 16 weeks.
- Placebo Comparator: Placebo + Letrozole: Participants received 2.5 mg letrozole tablets orally QD along with placebo on a 5-days-on/2-days-off schedule for a total of 16 weeks.
Period: Overall Study
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole
Started | 166 | 168
Completed | 157 | 160
Not Completed | 9 | 8
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Death | 1 | 0
Not completed — Non-compliance | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Progression of disease | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Reason not specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat (ITT) population includes all randomized participants regardless of whether they received any study drug (taselisib or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole | Total
Number analyzed (Participants) | 166 | 168 | 334
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (8.5) | 64.7 (8.7) | 64.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 168 | 334
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 143 | 140 | 283
  American Indian or Alaskan Native | 11 | 11 | 22
  Asian | 6 | 6 | 12
  Black or African American | 1 | 5 | 6
  Multiple | 1 | 0 | 1
  Other | 3 | 6 | 9
  Missing | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 48 | 84
  Not Hispanic or Latino | 114 | 109 | 223
  Not Reported | 13 | 10 | 23
  Unknown | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (OR) by Centrally Assessed Breast Magnetic Resonance Imaging (MRI) Via Modified Response Evaluation Criteria in Solid Tumors (mRECIST) Version 1.1
Description: Objective response rate (ORR) was defined as proportion of participants achieving complete response (CR) or partial response (PR). As per modified RECIST v1.1, CR: disappearance of all target lesions, PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: From Baseline to 16 weeks
Population: ITT population includes all randomized participants regardless of whether they received any study drug (taselisib or placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole
Number analyzed (Participants) | 166 | 168
percentage of participants | 50.0 | 39.3
Statistical Analysis 1: Comparison: Experimental: Taselisib + Letrozole vs Placebo Comparator: Placebo + Letrozole; Test type: Superiority; p = 0.0490, Cochran-Mantel-Haenszel; Difference in Response Rates = 10.71, 95% CI 2-sided [0.11 to 21.32]

2. Primary Outcome: Percentage of Participants With Total Pathologic Complete Response (Total pCR), Defined as Having pCR in Both Breast and Axilla, Using American Joint Committee on Cancer (AJCC) Staging System
Description: Total pCR was assessed by local pathology review on samples taken at surgery following completion of neoadjuvant therapy. tpCR was defined as the absence of any residual invasive cancer on hematoxylin and eosin evaluation of the resected breast specimen and all sampled ipsilateral lymph nodes ( i.e., ypT0/Tis, ypN0 in the AJCC staging system, 7th edition).
Time Frame: From Baseline to 16 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole
Number analyzed (Participants) | 166 | 168
percentage of participants | 1.8 | 0.6
Statistical Analysis 1: Comparison: Experimental: Taselisib + Letrozole vs Placebo Comparator: Placebo + Letrozole; Test type: Superiority; p = 0.3698, Fisher Exact; Difference in Response Rates = 1.21, 95% CI 2-sided [-1.12 to 3.55]

3. Primary Outcome: Percentage of Participants With OR by Centrally Assessed Breast MRI Via mRECIST Version 1.1 in Phosphatidylinositol-4,5-Bisphosphate 3-Kinase, Catalytic Subunit Alpha (PIK3CA) Mutant (MT) Participants
Description: ORR was defined as proportion of participants achieving CR or PR. As per modified RECIST v1.1, CR: disappearance of all target lesions, PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: From Baseline to 16 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole
Number analyzed (Participants) | 73 | 79
percentage of participants | 56.2 | 38.0
Statistical Analysis 1: Comparison: Experimental: Taselisib + Letrozole vs Placebo Comparator: Placebo + Letrozole; Test type: Superiority; p = 0.0332, Cochran-Mantel-Haenszel; Difference in Response Rates = 18.19, 95% CI 2-sided [2.57 to 33.81]

4. Primary Outcome: Percentage of Participants With Total pCR , Defined as Having pCR in Both Breast and Axilla, Using AJCC Staging System in PIK3CA MT Participants
Description: Total pCR was assessed by local pathology review on samples taken at surgery following completion of neoadjuvant therapy. tpCR was defined as the absence of any residual invasive cancer on hematoxylin and eosin evaluation of the resected breast specimen and all sampled ipsilateral lymph nodes (i.e., ypT0/Tis, ypN0 in the AJCC staging system, 7th edition).
Time Frame: From Baseline to 16 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole
Number analyzed (Participants) | 73 | 79
percentage of participants | 1.4 | 0
Statistical Analysis 1: Comparison: Experimental: Taselisib + Letrozole vs Placebo Comparator: Placebo + Letrozole; Test type: Superiority; p = 0.4803, Fisher Exact; Difference in Response Rates = 1.37, 95% CI 2-sided [-1.30 to 4.04]

5. Secondary Outcome: Percentage of Participants With OR by Centrally Assessed Breast MRI Via mRECIST Version 1.1 in PIK3CA Wildtype (WT) Participants
Description: as for outcome 3
Time Frame: From Baseline to 16 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole
Number analyzed (Participants) | 92 | 89
percentage of participants | 45.7 | 40.4
Statistical Analysis 1: Comparison: Experimental: Taselisib + Letrozole vs Placebo Comparator: Placebo + Letrozole; Test type: Superiority; p = 0.5017, Cochran-Mantel-Haenszel; Difference in Response Rates = 5.20, 95% CI 2-sided [-9.20 to 19.61]

6. Secondary Outcome: Percentage of Participants With Total pCR Defined as Having pCR in Both Breast and Axilla, Using AJCC Staging System in PIK3CA WT Participants
Description: as for outcome 4
Time Frame: From Baseline to 16 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole
Number analyzed (Participants) | 92 | 89
percentage of participants | 2.2 | 1.1
Statistical Analysis 1: Comparison: Experimental: Taselisib + Letrozole vs Placebo Comparator: Placebo + Letrozole; Test type: Superiority; p = 1.0000, Fisher Exact; Difference in Response Rates = 1.05, 95% CI 2-sided [-2.65 to 4.75]

7. Secondary Outcome: Percentage of Participants With OR by Breast Ultrasound Via mRECIST Version 1.1 in PIK3CA MT Participants
Description: as for outcome 3
Time Frame: From Baseline to 16 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole
Number analyzed (Participants) | 73 | 79
percentage of participants | 61.6 | 40.5
Statistical Analysis 1: Comparison: Experimental: Taselisib + Letrozole vs Placebo Comparator: Placebo + Letrozole; Test type: Superiority; p = 0.0115, Cochran-Mantel-Haenszel; Difference in Response Rates = 21.14, 95% CI 2-sided [5.59 to 36.68]

8. Secondary Outcome: Percentage of Participants With OR by Breast Ultrasound Via mRECIST Version 1.1 in PIK3CA WT Participants
Description: as for outcome 3
Time Frame: From Baseline to 16 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole
Number analyzed (Participants) | 92 | 89
percentage of participants | 54.3 | 51.7
Statistical Analysis 1: Comparison: Experimental: Taselisib + Letrozole vs Placebo Comparator: Placebo + Letrozole; Test type: Superiority; p = 0.7928, Cochran-Mantel-Haenszel; Difference in Response Rates = 2.66, 95% CI 2-sided [-11.88 to 17.20]

9. Secondary Outcome: Percentage of Participants With OR by Mammography Via mRECIST Version 1.1 in PIK3CA MT Participants
Description: as for outcome 3
Time Frame: From Baseline to 16 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole
Number analyzed (Participants) | 73 | 79
percentage of participants | 41.1 | 31.6
Statistical Analysis 1: Comparison: Experimental: Taselisib + Letrozole vs Placebo Comparator: Placebo + Letrozole; Test type: Superiority; p = 0.2659, Cochran-Mantel-Haenszel; Difference in Response Rates = 9.45, 95% CI 2-sided [-5.80 to 24.70]

10. Secondary Outcome: Percentage of Participants With OR by Mammography Via mRECIST Version 1.1 in PIK3CA WT Participants
Description: as for outcome 3
Time Frame: From Baseline to 16 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole
Number analyzed (Participants) | 92 | 89
percentage of participants | 40.2 | 32.6
Statistical Analysis 1: Comparison: Experimental: Taselisib + Letrozole vs Placebo Comparator: Placebo + Letrozole; Test type: Superiority; p = 0.3299, Cochran-Mantel-Haenszel; Difference in Response Rates = 7.63, 95% CI 2-sided [-6.34 to 21.60]

11. Secondary Outcome: Percentage of Participants With OR by Clinical Breast Exam (Palpation) Via mRECIST Version 1.1 in PIK3CA MT Participants
Description: as for outcome 3
Time Frame: From Baseline to 16 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole
Number analyzed (Participants) | 73 | 79
percentage of participants | 74.0 | 63.3
Statistical Analysis 1: Comparison: Experimental: Taselisib + Letrozole vs Placebo Comparator: Placebo + Letrozole; Test type: Superiority; p = 0.1554, Cochran-Mantel-Haenszel; Difference in Response Rates = 10.68, 95% CI 2-sided [-3.96 to 25.32]

12. Secondary Outcome: Percentage of Participants With OR by Clinical Breast Exam (Palpation) Via mRECIST Version 1.1 in PIK3CA WT Participants
Description: as for outcome 3
Time Frame: From Baseline to 16 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole
Number analyzed (Participants) | 92 | 89
percentage of participants | 62.0 | 59.6
Statistical Analysis 1: Comparison: Experimental: Taselisib + Letrozole vs Placebo Comparator: Placebo + Letrozole; Test type: Superiority; p = 0.7870, Cochran-Mantel-Haenszel; Difference in Response Rates = 2.41, 95% CI 2-sided [-11.82 to 16.63]

13. Secondary Outcome: Central Assessments of Changes in Ki67 Levels
Description: Ki67 is a prognostic marker and is used to evaluate the proliferative activity of breast cancer.
Time Frame: From Baseline to Week 3 and Surgery (Weeks 17-18); and Week 3 to Surgery (Weeks 17-18)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole
Number analyzed (Participants) | 166 | 168
percentage
  From Baseline to Week 3 | -83.81 [-86.73 to -80.23] | -80.44 [-83.93 to -76.19]
  From Baseline to Surgery | -75.58 [-80.45 to -69.49] | -80.51 [-84.41 to -75.64]
Statistical Analysis 1: Comparison: Experimental: Taselisib + Letrozole vs Placebo Comparator: Placebo + Letrozole; Statistical analysis for changes in Ki67 levels from Baseline to Week 3; Test type: Superiority; p = 0.117, Regression, Linear; Ratio of Least square mean = 0.83, 95% CI 2-sided [0.65 to 1.05]
Statistical Analysis 2: Comparison: Experimental: Taselisib + Letrozole vs Placebo Comparator: Placebo + Letrozole; Statistical analysis for changes in Ki67 levels from Baseline to Surgery; Test type: Superiority; p = 0.105, Regression, Linear; Ratio of Least square mean = 1.25, 95% CI 2-sided [0.95 to 1.65]

14. Secondary Outcome: Preoperative Endocrine Prognostic Index (PEPI ) Score
Description: To obtain the PEPI score, risk points for relapse-free survival (RFS) and breast cancer-specific survival (BCSS) are assigned depending on the hazard ratio (HR) from the multivariable analysis. The total PEPI score assigned to each participant is the sum of the risk points derived from the primary tumor (pT) stage, regional lymph nodes (pN) stage, Ki67 level, and estrogen receptor status of the surgical specimen. A HR in the range of 1 to 2 receives one risk point; a HR in the 2 to 2.5 range, two risk points; a HR greater than 2.5, three risk points. The total risk point score for each participant is the sum of all the risk points accumulated from the four factors in the model, ranges from 0 (best possible outcome) to 12 (worst possible outcome).
Time Frame: Week 16
Population: Data were not collected for this outcome measure.
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Percent Change From Baseline to Surgery in Enhancing Tumor Volume as Measured by Breast MRI
Time Frame: From Baseline to Surgery (Weeks 17-18)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percent change
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole
Number analyzed (Participants) | 166 | 168
percent change | -70.60 [-77.53 to -63.66] | -57.28 [-64.21 to -50.35]
Statistical Analysis 1: Comparison: Experimental: Taselisib + Letrozole vs Placebo Comparator: Placebo + Letrozole; Test type: Superiority; p = 0.002, Regression, Linear; Least squares mean difference = -13.32, 95% CI 2-sided [-21.67 to -4.96]

16. Secondary Outcome: Mean Score for Health-Related Quality of Life Measured by the European Organization for Research C30 (EORTC QLQ-C30)
Description: EORTC QLQ-C30 is a cancer-specific instrument with 30 questions used to assess the overall quality of life (QOL) in cancer participants. The first 28 questions used a 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much) for evaluating 5 functional scales (physical, role, social, cognitive, emotional), 8 symptom scales/items (diarrhea, fatigue, dyspnea, appetite loss, insomnia, nausea and vomiting [N/V], constipation, and pain) and a single item (financial difficulties). The last 2 questions represented the participant's assessment of overall health and quality of life, used 7-point scale (1=very poor to 7=excellent). EORTC QLQ-C30 global scores were linearly transformed on a scale of 0 to 100, with a high score indicating better QOL. Negative change from Baseline values indicated deterioration in QOL or functioning and positive values indicated improvement. Here, Post surgery= PS.
Time Frame: Weeks 1, 5, 9, 13, 16, 4-week Post-Surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole
Number analyzed (Participants) | 166 | 168
score on a scale
  Appetite Loss: Baseline: number analyzed (Participants) | 157 | 165
  Appetite Loss: Baseline | 6.2 (16.4) | 5.9 (14.2)
  Appetite Loss: Change at Week 5: number analyzed (Participants) | 155 | 160
  Appetite Loss: Change at Week 5 | 3.0 (18.4) | 1.9 (18.8)
  Appetite Loss: Change at Week 9: number analyzed (Participants) | 152 | 158
  Appetite Loss: Change at Week 9 | 5.3 (21.4) | 3.0 (17.8)
  Appetite Loss: Change at Week 13: number analyzed (Participants) | 152 | 157
  Appetite Loss: Change at Week 13 | 5.5 (23.8) | 2.1 (16.3)
  Appetite Loss: Change at Week 16: number analyzed (Participants) | 146 | 151
  Appetite Loss: Change at Week 16 | 6.8 (24.1) | 0.9 (16.3)
  Appetite Loss: Change at PS Visit: number analyzed (Participants) | 140 | 146
  Appetite Loss: Change at PS Visit | 5.0 (24.9) | 5.0 (23.3)
  Cognitive functioning: Baseline: number analyzed (Participants) | 158 | 163
  Cognitive functioning: Baseline | 90.8 (15.8) | 90.9 (16.6)
  Cognitive functioning: Change at Week 5: number analyzed (Participants) | 154 | 157
  Cognitive functioning: Change at Week 5 | 0.4 (12.8) | -2.5 (12.3)
  Cognitive functioning: Change at Week 9: number analyzed (Participants) | 151 | 157
  Cognitive functioning: Change at Week 9 | -1.1 (14.4) | -4.2 (14.7)
  Cognitive functioning: Change at Week 13: number analyzed (Participants) | 153 | 156
  Cognitive functioning: Change at Week 13 | -3.4 (15.8) | -5.1 (15.7)
  Cognitive functioning: Change at Week 16: number analyzed (Participants) | 147 | 147
  Cognitive functioning: Change at Week 16 | -4.2 (15.2) | -4.1 (17.5)
  Cognitive functioning: Change at PS Visit: number analyzed (Participants) | 140 | 144
  Cognitive functioning: Change at PS Visit | -3.1 (18.9) | -5.4 (16.8)
  Constipation: Baseline: number analyzed (Participants) | 158 | 164
  Constipation: Baseline | 6.8 (15.9) | 8.3 (18.2)
  Constipation: Change at Week 5: number analyzed (Participants) | 155 | 159
  Constipation: Change at Week 5 | 0.0 (16.1) | 3.1 (22.1)
  Constipation: Change at Week 9: number analyzed (Participants) | 151 | 158
  Constipation: Change at Week 9 | 0.2 (17.0) | 0.2 (18.6)
  Constipation: Change at Week 13: number analyzed (Participants) | 151 | 156
  Constipation: Change at Week 13 | -0.4 (18.5) | -0.6 (19.5)
  Constipation: Change at Week 16: number analyzed (Participants) | 146 | 148
  Constipation: Change at Week 16 | -1.1 (17.2) | 1.6 (20.3)
  Constipation: Change at PS Visit: number analyzed (Participants) | 140 | 145
  Constipation: Change at PS Visit | 4.8 (23.2) | 1.1 (16.9)
  Diarrhoea: Baseline: number analyzed (Participants) | 157 | 163
  Diarrhoea: Baseline | 5.9 (14.9) | 4.3 (11.8)
  Diarrhoea: Change at Week 5: number analyzed (Participants) | 154 | 155
  Diarrhoea: Change at Week 5 | 6.7 (21.7) | -0.2 (13.4)
  Diarrhoea: Change at Week 9: number analyzed (Participants) | 150 | 157
  Diarrhoea: Change at Week 9 | 6.4 (24.3) | 0.8 (15.1)
  Diarrhoea: Change at Week 13: number analyzed (Participants) | 152 | 155
  Diarrhoea: Change at Week 13 | 7.9 (22.3) | -0.4 (14.7)
  Diarrhoea: Change at Week 16: number analyzed (Participants) | 146 | 146
  Diarrhoea: Change at Week 16 | 8.4 (23.1) | 0.2 (16.4)
  Diarrhoea: Change at PS Visit: number analyzed (Participants) | 140 | 144
  Diarrhoea: Change at PS Visit | 0.2 (17.7) | -0.9 (15.7)
  Dyspnoea: Baseline: number analyzed (Participants) | 157 | 165
  Dyspnoea: Baseline | 7.4 (15.8) | 8.5 (17.5)
  Dyspnoea: Change at Week 5: number analyzed (Participants) | 154 | 160
  Dyspnoea: Change at Week 5 | -0.2 (14.0) | 0.6 (18.1)
  Dyspnoea: Change at Week 9: number analyzed (Participants) | 150 | 159
  Dyspnoea: Change at Week 9 | 2.0 (17.4) | 1.9 (19.9)
  Dyspnoea: Change at Week 13: number analyzed (Participants) | 151 | 157
  Dyspnoea: Change at Week 13 | 3.5 (21.1) | 1.7 (22.3)
  Dyspnoea: Change at Week 16: number analyzed (Participants) | 146 | 151
  Dyspnoea: Change at Week 16 | 3.4 (20.2) | 2.6 (22.6)
  Dyspnoea: Change at PS Visit: number analyzed (Participants) | 138 | 146
  Dyspnoea: Change at PS Visit | 3.1 (24.8) | 2.1 (21.5)
  Emotional functioning: Baseline: number analyzed (Participants) | 158 | 163
  Emotional functioning: Baseline | 77.0 (20.4) | 78.2 (19.9)
  Emotional functioning: Change at Week 5: number analyzed (Participants) | 154 | 157
  Emotional functioning: Change at Week 5 | 4.2 (15.2) | 2.4 (17.0)
  Emotional functioning: Change at Week 9: number analyzed (Participants) | 151 | 157
  Emotional functioning: Change at Week 9 | 3.8 (14.7) | 1.3 (20.7)
  Emotional functioning: Change at Week 13: number analyzed (Participants) | 153 | 156
  Emotional functioning: Change at Week 13 | 2.5 (15.2) | -1.4 (18.6)
  Emotional functioning: Change at Week 16: number analyzed (Participants) | 147 | 147
  Emotional functioning: Change at Week 16 | 1.0 (17.0) | -3.5 (20.2)
  Emotional functioning: Change at PS Visit: number analyzed (Participants) | 140 | 144
  Emotional functioning: Change at PS Visit | -0.8 (19.0) | -3.6 (20.9)
  Fatigue: Baseline: number analyzed (Participants) | 158 | 165
  Fatigue: Baseline | 14.8 (18.7) | 15.6 (18.5)
  Fatigue: Change at Week 5: number analyzed (Participants) | 155 | 161
  Fatigue: Change at Week 5 | 4.7 (13.9) | 4.9 (17.9)
  Fatigue: Change at Week 9: number analyzed (Participants) | 152 | 159
  Fatigue: Change at Week 9 | 5.0 (15.9) | 7.5 (20.3)
  Fatigue: Change at Week 13: number analyzed (Participants) | 151 | 158
  Fatigue: Change at Week 13 | 7.9 (18.1) | 8.8 (21.4)
  Fatigue: Change at Week 16: number analyzed (Participants) | 146 | 151
  Fatigue: Change at Week 16 | 6.8 (17.5) | 8.0 (20.4)
  Fatigue: Change at PS Visit: number analyzed (Participants) | 140 | 146
  Fatigue: Change at PS Visit | 12.3 (19.5) | 12.4 (22.6)
  Financial difficulties: Baseline: number analyzed (Participants) | 156 | 160
  Financial difficulties: Baseline | 9.0 (20.9) | 10.0 (20.4)
  Financial difficulties: Change at Week 5: number analyzed (Participants) | 152 | 154
  Financial difficulties: Change at Week 5 | -2.6 (14.6) | -0.4 (20.2)
  Financial difficulties: Change at Week 9: number analyzed (Participants) | 151 | 153
  Financial difficulties: Change at Week 9 | -2.6 (17.9) | 0.7 (20.4)
  Financial difficulties: Change at Week 13: number analyzed (Participants) | 150 | 152
  Financial difficulties: Change at Week 13 | -1.1 (17.9) | 0.0 (19.9)
  Financial difficulties: Change at Week 16: number analyzed (Participants) | 145 | 144
  Financial difficulties: Change at Week 16 | -1.1 (15.9) | 2.1 (24.4)
  Financial difficulties: Change at PS Visit: number analyzed (Participants) | 138 | 141
  Financial difficulties: Change at PS Visit | 1.9 (20.0) | 3.8 (23.6)
  Global health status / QoL: Baseline: number analyzed (Participants) | 158 | 162
  Global health status / QoL: Baseline | 75.3 (19.7) | 74.6 (21.2)
  Global health status / QoL: Change at Week 5: number analyzed (Participants) | 153 | 156
  Global health status / QoL: Change at Week 5 | 1.5 (15.2) | -1.1 (18.5)
  Global health status / QoL: Change at Week 9: number analyzed (Participants) | 150 | 155
  Global health status / QoL: Change at Week 9 | -1.1 (15.9) | -3.2 (22.7)
  Global health status / QoL: Change at Week 13: number analyzed (Participants) | 152 | 155
  Global health status / QoL: Change at Week 13 | -2.4 (19.5) | -3.7 (20.7)
  Global health status / QoL: Change at Week 16: number analyzed (Participants) | 147 | 146
  Global health status / QoL: Change at Week 16 | -2.2 (18.4) | -2.9 (22.6)
  Global health status / QoL: Change at PS Visit: number analyzed (Participants) | 139 | 143
  Global health status / QoL: Change at PS Visit | -5.9 (19.7) | -7.0 (22.2)
  Insomnia: Baseline: number analyzed (Participants) | 158 | 165
  Insomnia: Baseline | 23.0 (27.1) | 22.4 (28.1)
  Insomnia: Change at Week 5: number analyzed (Participants) | 155 | 161
  Insomnia: Change at Week 5 | -2.4 (24.1) | -0.4 (27.6)
  Insomnia: Change at Week 9: number analyzed (Participants) | 151 | 159
  Insomnia: Change at Week 9 | -1.8 (24.9) | -0.6 (26.9)
  Insomnia: Change at Week 13: number analyzed (Participants) | 153 | 158
  Insomnia: Change at Week 13 | -1.1 (27.7) | 2.1 (29.5)
  Insomnia: Change at Week 16: number analyzed (Participants) | 146 | 149
  Insomnia: Change at Week 16 | -0.7 (26.1) | -2.2 (27.6)
  Insomnia: Change at PS Visit: number analyzed (Participants) | 140 | 146
  Insomnia: Change at PS Visit | -1.4 (26.8) | 3.2 (34.4)
  Nausea and vomiting: Baseline: number analyzed (Participants) | 158 | 165
  Nausea and vomiting: Baseline | 1.9 (7.5) | 1.6 (6.2)
  Nausea and vomiting: Change at Week 5: number analyzed (Participants) | 155 | 161
  Nausea and vomiting: Change at Week 5 | 3.7 (11.3) | 1.9 (9.9)
  Nausea and vomiting: Change at Week 9: number analyzed (Participants) | 152 | 159
  Nausea and vomiting: Change at Week 9 | 3.4 (10.9) | 1.7 (10.3)
  Nausea and vomiting: Change at Week 13: number analyzed (Participants) | 153 | 158
  Nausea and vomiting: Change at Week 13 | 3.7 (12.9) | 0.7 (8.5)
  Nausea and vomiting: Change at Week 16: number analyzed (Participants) | 146 | 151
  Nausea and vomiting: Change at Week 16 | 2.5 (14.0) | 0.6 (8.0)
  Nausea and vomiting: Change at PS Visit: number analyzed (Participants) | 140 | 146
  Nausea and vomiting: Change at PS Visit | 2.1 (14.8) | 1.0 (8.6)
  Pain: Baseline: number analyzed (Participants) | 157 | 165
  Pain: Baseline | 13.1 (20.4) | 12.3 (19.6)
  Pain: Change at Week 5: number analyzed (Participants) | 155 | 161
  Pain: Change at Week 5 | -0.6 (18.8) | 2.6 (17.5)
  Pain: Change at Week 9: number analyzed (Participants) | 152 | 159
  Pain: Change at Week 9 | -1.8 (16.5) | 3.8 (22.9)
  Pain: Change at Week 13: number analyzed (Participants) | 152 | 158
  Pain: Change at Week 13 | -1.4 (18.4) | 4.7 (23.4)
  Pain: Change at Week 16: number analyzed (Participants) | 147 | 151
  Pain: Change at Week 16 | -0.9 (19.1) | 1.8 (22.0)
  Pain: Change at PS Visit: number analyzed (Participants) | 140 | 146
  Pain: Change at PS Visit | 11.1 (26.0) | 13.8 (26.6)
  Physical functioning: Baseline: number analyzed (Participants) | 158 | 165
  Physical functioning: Baseline | 89.6 (13.7) | 90.8 (13.4)
  Physical functioning: Change at Week 5: number analyzed (Participants) | 155 | 161
  Physical functioning: Change at Week 5 | 0.5 (9.6) | -1.2 (11.5)
  Physical functioning: Change at Week 9: number analyzed (Participants) | 152 | 157
  Physical functioning: Change at Week 9 | 0.2 (10.1) | -2.0 (13.1)
  Physical functioning: Change at Week 13: number analyzed (Participants) | 152 | 158
  Physical functioning: Change at Week 13 | -0.3 (12.4) | -1.9 (14.0)
  Physical functioning: Change at Week 16: number analyzed (Participants) | 146 | 150
  Physical functioning: Change at Week 16 | -0.5 (10.9) | -3.4 (15.1)
  Physical functioning: Change at PS Visit: number analyzed (Participants) | 140 | 146
  Physical functioning: Change at PS Visit | -5.2 (16.0) | -7.5 (15.7)
  Role functioning: Baseline: number analyzed (Participants) | 157 | 165
  Role functioning: Baseline | 90.7 (20.1) | 93.1 (16.5)
  Role functioning:Change at Week 5: number analyzed (Participants) | 155 | 160
  Role functioning:Change at Week 5 | 1.3 (14.3) | -2.5 (17.1)
  Role functioning:Change at Week 9: number analyzed (Participants) | 150 | 159
  Role functioning:Change at Week 9 | -0.2 (12.8) | -4.9 (18.9)
  Role functioning:Change at Week 13: number analyzed (Participants) | 152 | 157
  Role functioning:Change at Week 13 | -2.3 (17.4) | -5.6 (19.8)
  Role functioning:Change at Week 16: number analyzed (Participants) | 146 | 151
  Role functioning:Change at Week 16 | -4.6 (16.3) | -4.4 (18.9)
  Role functioning:Change at PS Visit: number analyzed (Participants) | 140 | 146
  Role functioning:Change at PS Visit | -15.1 (24.7) | -20.1 (28.1)
  Social functioning: Baseline: number analyzed (Participants) | 155 | 161
  Social functioning: Baseline | 91.2 (17.6) | 94.9 (14.3)
  Social functioning: Change at Week 5: number analyzed (Participants) | 151 | 155
  Social functioning: Change at Week 5 | 3.1 (12.8) | -2.0 (15.7)
  Social functioning: Change at Week 9: number analyzed (Participants) | 150 | 155
  Social functioning: Change at Week 9 | 2.0 (13.4) | -4.0 (18.1)
  Social functioning: Change at Week 13: number analyzed (Participants) | 150 | 154
  Social functioning: Change at Week 13 | 0.0 (13.7) | -4.0 (19.0)
  Social functioning: Change at Week 16: number analyzed (Participants) | 146 | 145
  Social functioning: Change at Week 16 | -0.5 (13.7) | -3.1 (19.3)
  Social functioning: Change at PS Visit: number analyzed (Participants) | 139 | 142
  Social functioning: Change at PS Visit | -6.4 (20.3) | -10.1 (24.2)

17. Secondary Outcome: Mean Score for Treatment of Cancer Quality of Life Questionnaire BR23 (QLQ-BR23)
Description: EORTC-QLQ-BR23 is a 23-item breast cancer-specific companion module to the EORTC-QLQ-C30 and consists of four functional scales (body image, sexual enjoyment, sexual functioning, future perspective [FP]) and four symptom scales (systemic side effects [SE], upset by hair loss, arm symptoms, breast symptoms). Questions used 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Scores were averaged and transformed to 0-100 scale. High score for functional scale indicated high/better level of functioning/healthy functioning. Negative change from Baseline indicated deterioration in QOL and positive change from Baseline indicated an improvement in QOL. Here, Post surgery= PS.
Time Frame: Weeks 1, 5, 9, 13, 16, 4-week Post-Surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole
Number analyzed (Participants) | 166 | 168
score on a scale
  Body image: Baseline: number analyzed (Participants) | 155 | 160
  Body image: Baseline | 91.8 (15.7) | 94.0 (14.6)
  Body image: Change at Week 5: number analyzed (Participants) | 152 | 151
  Body image: Change at Week 5 | 2.8 (8.8) | 0.6 (11.4)
  Body image: Change at Week 9: number analyzed (Participants) | 149 | 150
  Body image: Change at Week 9 | 1.2 (9.8) | -0.2 (10.3)
  Body image: Change at Week 13: number analyzed (Participants) | 150 | 149
  Body image: Change at Week 13 | 1.2 (11.6) | -1.6 (13.8)
  Body image: Change at Week 16: number analyzed (Participants) | 145 | 143
  Body image: Change at Week 16 | 0.1 (10.8) | -1.2 (12.8)
  Body image: Change at PS Visit: number analyzed (Participants) | 138 | 140
  Body image: Change at PS Visit | -6.5 (22.3) | -8.3 (19.2)
  Breast symptoms: Baseline: number analyzed (Participants) | 154 | 160
  Breast symptoms: Baseline | 5.3 (9.8) | 6.9 (12.7)
  Breast symptoms: Change at Week 5: number analyzed (Participants) | 148 | 150
  Breast symptoms: Change at Week 5 | 2.3 (14.6) | 1.0 (13.0)
  Breast symptoms: Change at Week 9: number analyzed (Participants) | 148 | 151
  Breast symptoms: Change at Week 9 | 4.5 (15.1) | 1.8 (11.7)
  Breast symptoms: Change at Week 13: number analyzed (Participants) | 149 | 151
  Breast symptoms: Change at Week 13 | 5.8 (16.0) | 2.3 (13.3)
  Breast symptoms: Change at Week 16: number analyzed (Participants) | 146 | 146
  Breast symptoms: Change at Week 16 | 7.9 (18.6) | 3.9 (14.9)
  Breast symptoms: Change at PS Visit: number analyzed (Participants) | 136 | 140
  Breast symptoms: Change at PS Visit | 6.6 (17.9) | 4.3 (14.2)
  Future perspective: Baseline: number analyzed (Participants) | 157 | 159
  Future perspective: Baseline | 57.7 (31.0) | 58.7 (29.9)
  Future perspective: Change at Week 5: number analyzed (Participants) | 154 | 151
  Future perspective: Change at Week 5 | 6.5 (26.7) | 9.3 (28.1)
  Future perspective: Change at Week 9: number analyzed (Participants) | 150 | 151
  Future perspective: Change at Week 9 | 10.2 (25.0) | 9.7 (26.6)
  Future perspective: Change at Week 13: number analyzed (Participants) | 151 | 152
  Future perspective: Change at Week 13 | 7.7 (28.4) | 4.4 (29.1)
  Future perspective: Change at Week 16: number analyzed (Participants) | 147 | 145
  Future perspective: Change at Week 16 | 10.2 (26.1) | 5.1 (29.2)
  Future perspective: Change at PS Visit: number analyzed (Participants) | 139 | 139
  Future perspective: Change at PS Visit | 6.5 (29.7) | 3.4 (34.8)
  Sexual enjoyment: Baseline: number analyzed (Participants) | 48 | 29
  Sexual enjoyment: Baseline | 41.7 (22.3) | 47.1 (28.9)
  Sexual enjoyment: Change at Week 5: number analyzed (Participants) | 40 | 24
  Sexual enjoyment: Change at Week 5 | 3.3 (18.2) | 11.1 (23.4)
  Sexual enjoyment: Change at Week 9: number analyzed (Participants) | 40 | 22
  Sexual enjoyment: Change at Week 9 | 8.3 (23.6) | 10.6 (23.9)
  Sexual enjoyment: Change at Week 13: number analyzed (Participants) | 33 | 21
  Sexual enjoyment: Change at Week 13 | 6.1 (19.5) | 1.6 (22.3)
  Sexual enjoyment: Change at Week 16: number analyzed (Participants) | 34 | 22
  Sexual enjoyment: Change at Week 16 | 9.8 (19.3) | 7.6 (22.8)
  Sexual enjoyment: Change at PS Visit: number analyzed (Participants) | 21 | 15
  Sexual enjoyment: Change at PS Visit | 14.3 (27.0) | 2.2 (23.5)
  Sexual functioning: Baseline: number analyzed (Participants) | 149 | 147
  Sexual functioning: Baseline | 81.2 (23.4) | 85.1 (20.2)
  Sexual functioning: Change at Week 5: number analyzed (Participants) | 144 | 133
  Sexual functioning: Change at Week 5 | 1.2 (13.6) | 1.0 (15.0)
  Sexual functioning: Change at Week 9: number analyzed (Participants) | 136 | 131
  Sexual functioning: Change at Week 9 | 1.3 (14.5) | 0.3 (16.5)
  Sexual functioning: Change at Week 13: number analyzed (Participants) | 129 | 126
  Sexual functioning: Change at Week 13 | 4.1 (16.1) | 1.6 (17.7)
  Sexual functioning: Change at Week 16: number analyzed (Participants) | 128 | 124
  Sexual functioning: Change at Week 16 | 4.8 (15.9) | 1.1 (18.1)
  Sexual functioning: Change at PS Visit: number analyzed (Participants) | 120 | 121
  Sexual functioning: Change at PS Visit | 9.6 (19.2) | 4.1 (21.8)
  Systematic therapy side effects: Baseline: number analyzed (Participants) | 159 | 162
  Systematic therapy side effects: Baseline | 8.7 (10.8) | 9.5 (11.5)
  Systematic therapy side effects: Change at Week 5: number analyzed (Participants) | 156 | 153
  Systematic therapy side effects: Change at Week 5 | 4.3 (10.0) | 3.9 (10.5)
  Systematic therapy side effects: Change at Week 9: number analyzed (Participants) | 153 | 154
  Systematic therapy side effects: Change at Week 9 | 6.7 (10.8) | 5.9 (12.1)
  Systematic therapy side effects: Change at Week 13: number analyzed (Participants) | 154 | 155
  Systematic therapy side effects: Change at Week 13 | 7.3 (11.0) | 6.2 (13.1)
  Systematic therapy side effects: Change at Week 16: number analyzed (Participants) | 149 | 149
  Systematic therapy side effects: Change at Week 16 | 7.5 (12.9) | 7.1 (12.6)
  Systematic therapy side effects:Change at PS Visit: number analyzed (Participants) | 141 | 142
  Systematic therapy side effects:Change at PS Visit | 7.0 (12.0) | 5.9 (12.1)
  Upset by hair loss: Baseline: number analyzed (Participants) | 19 | 18
  Upset by hair loss: Baseline | 24.6 (26.9) | 35.2 (31.3)
  Upset by hair loss: Change at Week 5: number analyzed (Participants) | 12 | 10
  Upset by hair loss: Change at Week 5 | 11.1 (32.8) | -3.3 (18.9)
  Upset by hair loss: Change at Week 9: number analyzed (Participants) | 11 | 11
  Upset by hair loss: Change at Week 9 | 9.1 (44.9) | -9.1 (26.2)
  Upset by hair loss: Change at Week 13: number analyzed (Participants) | 10 | 11
  Upset by hair loss: Change at Week 13 | 16.7 (36.0) | -3.0 (34.8)
  Upset by hair loss: Change at Week 16: number analyzed (Participants) | 11 | 14
  Upset by hair loss: Change at Week 16 | 21.2 (34.2) | -7.1 (23.3)
  Upset by hair loss: Change at PS Visit: number analyzed (Participants) | 13 | 13
  Upset by hair loss: Change at PS Visit | 30.8 (37.2) | -2.6 (34.6)

18. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Baseline up to 22 weeks
Population: The safety population includes all randomized participants who received at least one dose of taselisib or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole
Number analyzed (Participants) | 167 | 167
percentage of participants | 91.0 | 83.2

ADVERSE EVENTS:
Time Frame: Baseline up to 22 weeks
Description: The safety population includes all randomized participants who received at least one dose of taselisib or placebo.
Arm/Group | Experimental: Taselisib + Letrozole | Placebo Comparator: Placebo + Letrozole
All-Cause Mortality (participants affected / at risk) | 1/167 | 0/167
Serious Adverse Events (participants affected / at risk) | 20/167 | 4/167
Other Adverse Events (participants affected / at risk) | 130/167 | 126/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Taselisib + Letrozole (N=167) | Placebo Comparator: Placebo + Letrozole (N=167)
Postoperative wound infection (Infections and infestations) | 2 | 1
Erysipelas (Infections and infestations) | 2 | 0
Bacterial diarrhoea (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 0
Colitis (Gastrointestinal disorders) | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Taselisib + Letrozole (N=167) | Placebo Comparator: Placebo + Letrozole (N=167)
Diarrhoea (Gastrointestinal disorders) | 49 | 20
Nausea (Gastrointestinal disorders) | 35 | 19
Stomatitis (Gastrointestinal disorders) | 22 | 5
Dry mouth (Gastrointestinal disorders) | 6 | 14
Constipation (Gastrointestinal disorders) | 10 | 7
Vomiting (Gastrointestinal disorders) | 10 | 6
Dyspepsia (Gastrointestinal disorders) | 9 | 1
Fatigue (General disorders) | 33 | 40
Asthenia (General disorders) | 17 | 16
Viral upper respiratory tract infection (Infections and infestations) | 6 | 13
Urinary tract infection (Infections and infestations) | 7 | 9
Alanine aminotransferase increased (Investigations) | 9 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 26 | 12
Decreased appetite (Metabolism and nutrition disorders) | 11 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 36
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 10
Headache (Nervous system disorders) | 16 | 18
Dizziness (Nervous system disorders) | 9 | 9
Insomnia (Psychiatric disorders) | 6 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 8
Rash (Skin and subcutaneous tissue disorders) | 15 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 3
Hot flush (Vascular disorders) | 25 | 33
Hypertension (Vascular disorders) | 10 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2015-07-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT02273973/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT02273973/SAP_001.pdf